CLINICAL TRIAL: NCT04512456
Title: Autonomic and Hemodynamic Responses to Muscular Ergoreflex Activation in People Living With HIV/AIDS: Effects of Exercise Training.
Brief Title: Cardiovascular Responses to Exercise in People Living With HIV/AIDS: Effects of Exercise Training
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Cardiologia de Laranjeiras (Other)
Collaborators: Rio de Janeiro State University (Other)
Responsible Party: Principal Investigator, Juliana Pereira Borges, Professor, Rio de Janeiro State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: FAPERJ E-26/010.100935/2018
Record Dates: First submitted 2020-08-07; First posted 2020-08-13 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: HIV+active group will perform exercise training, while HIV+inactive and HIV- groups will not undergo intervention.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Active HIV-infected patients (Experimental): Exercise training
  Interventions: Behavioral: Exercise training
- Inactive HIV-infected patients (No Intervention): No intervention.
- Healthy subjects (No Intervention): No intervention.

INTERVENTIONS:
Behavioral: Exercise training — Exercise training performed during 12 weeks, 3 sessions per week of 60 minutes of strength and aerobic exercises.
  Arms: Active HIV-infected patients

SUMMARY:
Patients living with HIV (PLWHIV) have compromised muscle metaboreflex, which can cause exercise intolerance. This randomized controlled clinical trial will verify the effects of regular exercise on autonomic and hemodynamic responses to muscle ergoreflex activation in these patients. PLWHIV without regular physical exercise will be randomly assigned into an exercise training or a control group. The exercise training group will undergo regular physical exercise during 12 weeks (60-min session performed 3 times/wk with moderate intensity), while the control group will keep inactive. Another group consisted of inactive HIV-uninfected group will be included. The primary endpoints will be blood pressure and autonomic markers in response to the Stroop Color-Word Test and the activation of muscle ergoreflex, by means of the post-exercise circulatory arrest (PECA), which will be performed with and without the topical application of a capsaicin-based analgesic balm. Secondary endpoints will include heart rate, peripheral vascular resistance, stroke volume, cardiac output, blood lactate concentration, anthropometrics, and handgrip strength. The active and inactive PLWHIV groups will be evaluated before and after the exercise training, while the healthy group only at baseline.

DETAILED DESCRIPTION:
HIV-infection is associated to a reduced maximal cardiac output and blunted pressor reflex response to static handgrip exercise, which are suggestive of impaired ergoreflex activation. An abnormal ergoreflex activation may lead to exercise intolerance and increases in cardiovascular risk. Despite the importance of therapeutic strategies in reducing the cardiovascular risk among patients living with HIV, exercise-related effects on ergoreflex sensitivity in these population have not been previously investigated.

ELIGIBILITY:
Inclusion Criteria for people living with HIV:

* diagnosis of HIv infection for at least 5 years;
* use of combined antiretroviral therapy for at least 3 years;
* asymptomatic and free from opportunistic diseases at enrollment.

Exclusion Criteria:

* regular physical exercise;
* malnutrition;
* presence of coronary artery disease, ischemic diseases, pulmonary disease, diabetes, Chagas disease, tuberculosis, heart failure, hypertension;
* using pacemakers and/or antidepressant, antiarrhythmic or antihypertensive medication, especially beta-blockers.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Blood Pressure at 3 months | Baseline and 3 months of follow-up
  Blood pressure will be assessed by a digital sphygmomanometer.
Change from Baseline Heart Rate Variability at 3 months | Baseline and 3 months of follow-up
  Heart rate variability will be assessed by a heart rate monitor.

SECONDARY OUTCOMES:
Change from Baseline Heart Rate at 3 months | Baseline and 3 months of follow-up
  Heart rate will be evaluated beat-to-beat by means of a heart rate monitor.
Change from Baseline Peripheral Vascular Resistance at 3 months | Baseline and 3 months of follow-up
  Peripheral Vascular Resistance will be evaluated by photpletismography.
Change from Baseline Stroke Volume at 3 months | Baseline and 3 months of follow-up
  Stroke Volume will be evaluated by photoplethysmography.
Change from Baseline Cardiac Output at 3 months | Baseline and 3 months of follow-up
  Cardiac Output will be evaluated by photoplethysmography.
Change from Baseline Blood Lactate at 3 months | Baseline and 3 months of follow-up.
  Blood Lactate will be determined by the YSL 2700 analyzer.
Change from Baseline Anthropometric markers at 3 months | Baseline and 3 months of follow-up.
  Anthropometric markers will be determined by a digital scale and wall-mounted stadiometer.
Change from Baseline handgrip maximal voluntary contraction at 3 months | Baseline and 3 months of follow-up.
  Handgrip maximal voluntary contraction will be assessed using a hydraulic handgrip dynamometer.

CONTACTS AND LOCATIONS:
Overall Officials: Julana P Borges, Dr, Principal Investigator — Rio de Janeiro State University
Locations (1):
- Rio de Janeiro State University, Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gama G, Dos Santos Rangel MV, de Oliveira Coelho VC, Paz GA, de Matos CVB, Silva BP, Lopes GO, Lopes KG, Farinatti P, Borges JP. The effects of exercise training on autonomic and hemodynamic responses to muscle metaboreflex in people living with HIV/AIDS: A randomized clinical trial protocol. PLoS One. 2022 Mar 18;17(3):e0265516. doi: 10.1371/journal.pone.0265516. eCollection 2022. PMID 35303017